CLINICAL TRIAL: NCT05479136
Title: 18F-Fluciclovine PET Imaging for Detecting High Grade Glioma Recurrence After Radiochemotherapy
Acronym: DRARCH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nicole Hill (Other)
Collaborators: Blue Earth Diagnostics (Industry); Barrow Neurological Foundation (Other)
Responsible Party: Sponsor-Investigator, Nicole Hill, Program Manager, St. Joseph's Hospital and Medical Center, Phoenix
Organization: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PHX-22-500-229-30-08; BED-IIT-420 (Other: Blue Earth Diagnostics)
Record Dates: First submitted 2022-06-24; First posted 2022-07-29 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-10

CONDITIONS: Grade III or Grade IV Glioma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — Magnetic Resonance Spectroscopy; fluciclovine F-18

STUDY DESIGN:
Intervention Model Description: Up to 30 eligible patients will be recruited from out-patient clinic visits at Barrow Neurological Institute.
Masking Description: All participants will receive the same imaging.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- PET study (Experimental): Single intravenous administration of 18F fluciclovine for PET Scan
  Interventions: Drug: PET imaging with 18F fluciclovine

INTERVENTIONS:
Drug: PET imaging with 18F fluciclovine — PET with 18F fluciclovine injection, 185 MBq (5 mCi) ± 20%, delivered as an intravenous bolus
  Other Names: Axumin

SUMMARY:
This study will examine whether positron emission tomography (PET) imaging with fluciclovine can reliably differentiate true progression from pseudoprogression months earlier than the conventional MRI methods.

DETAILED DESCRIPTION:
Approximately 40-50% of all glioblastoma patients undergoing standard of care radiochemotherapy will show signs of early disease progression that includes increases in the apparent tumor size on conventional magnetic resonance imaging (MRI) scans. Unfortunately, treatment related effects, including alterations to the blood brain barrier (BBB), can mimic tumor progression on conventional MRI scans, which confounds assessment of tumor progression during and in the months following radiochemotherapy.

An imaging method that provides a reliable early assessment of brain tumor progression could enable patients to enroll into clinical trials months earlier (when tumors are more treatable) and potentially save patients from the adverse side effects of an ineffective radiochemotherapy regimen. Fluciclovine positron emission tomography (PET) imaging has the potential to overcome the limitations of conventional MRI and provide an earlier, more comprehensive assessment of brain tumor progression. Fluciclovine is a radiolabeled amino acid analogue whose transport across the BBB and retention in tumor cells is dictated primarily by upregulated amino acid transporters. Prior studies have shown that amino acid PET with radiotracers similar to fluciclovine can accurately distinguish tumor progression from treatment effects in glioma patients, but these other amino acid radiotracers are not widely available. Another advantage of fluciclovine PET is that is can detect infiltrative tumor cells that are often not discernable on standard conventional MRI and are often in regions beyond that those with disrupted BBB. There are no published studies evaluating whether fluciclovine PET can differentiate progression from treatment effects despite fluciclovine being commercially available and widely accessible. The goals of this proposal are to establish whether fluciclovine PET can: i) identify early progression at time points soon after completion of radiation therapy and ii) differentiate treatment-related effects from true disease progression in patients with suspected recurrent disease.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than 18 years of age
2. Histological diagnosis of primary WHO grade III or IV glioma
3. Completed standard radiotherapy
4. Undergoing or completed standard chemotherapy (or other therapies)
5. Enlarging or new contrast-enhancing mass suspicious for progression/recurrence (at least 10mm in one direction)
6. Subjects must agree to take adequate pregnancy preventions from the time of consent until 24 hrs after the 18F-fluciclovine injection.
7. Willing and able to provide written informed consent in compliance with the regulatory requirements. If a subject is unable to provide written informed consent, written informed consent may be obtained from the subject's legal representative

Exclusion Criteria:

1. Simultaneous participation in other interventional trials which could interfere with this trial.
2. Inability to undergo a MRI or PET scan (claustrophobia, non-MRI compatible pacemaker, renal insufficiency, known allergy to MRI contrast agent or fluciclovine tracer)
3. Subjects who are pregnant or lactating or who suspect they might be pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-24 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Brain tumor progression | 20 weeks
  whether fluciclovine PET, a commercially available tracer, provides A reliable measure of brain tumor progression months earlier than conventional MRI.

SECONDARY OUTCOMES:
PET uptake and dynamic susceptibility contrast (DSC) perfusion | 20 weeks
  Establish the spatial correlation between PET uptake and dynamic susceptibility contrast (DSC) perfusion MRI measurements of relative cerebral blood volume (rCBV).

CONTACTS AND LOCATIONS:
Overall Officials: Poonam Choudhary, PhD, Principal Investigator — Barrow Neurological Institute
Locations (1):
- Barrow Neurological Institute at St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No